CLINICAL TRIAL: NCT06903507
Title: The Comfort Study: Determining the Most Comfortable Radiotherapy Mattress
Brief Title: Increasing Patient Comfort in Palliative Radiotherapy With a Newly Developed Mattress - A Prospective Clinical Study
Acronym: RTCOMFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Royal Health Foam (Unknown)
Responsible Party: Principal Investigator, Steven Petit, Associate Professor, Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2023-0295
Record Dates: First submitted 2025-03-21; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms
Keywords: radiotherapy; palliative radiotherapy; radiation oncology; comfort; pain; mattress; bone metastasis
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT-Comfort Mattress (Experimental): In this arm, the RT-Comfort Mattress was applied on top of the flat and hard radiotherapy treatment couch during planning CT acquisition and treatment dose delivery.
  Interventions: Device: RT-Comfort Mattress
- Standard thin foam matt (No Intervention): For patients with painful bone metastasis, a standard thin foam matt is typically added on top of the flat and hard radiotherapy treatment couch to somewhat relief the pain. Unfortunately, this existing matt is too thin to effectively counter discomfort and pain.

INTERVENTIONS:
Device: RT-Comfort Mattress — This dedicated RT-Comfort Mattress was newly developed (patent pending) for increasing comfort without compromising radiotherapy treatment quality.
  Arms: RT-Comfort Mattress

SUMMARY:
The goal of this research is to determine if a new radiotherapy mattress is more comfortable for patients than the standard mattress. The table of the CT scanner and the radiation machine is flat and hard. To increase comfort during the CT scan and radiation dose delivery, the investigators have recently developed a new mattress (RTComfort). This research aims to find out if the new mattress is more comfortable for patients than the standard matt and to learn how radiotherapy mattresses can be further improved.

Patients who participate in the research, will be asked to try both the standard mattress and the new mattress during the CT scan appointment. This will take about 5 minutes (one minute each). Patients will then be asked which mattress was most comfortable and if they experience any pain while lying on the mattress. Patients can choose which mattress will be used for the CT scan and treatment. Both mattresses are approved and safe for treatment. If patients participate in the research, it means the investigators will collect and use some of their (medical) data.

Patients will not have any direct benefits from participating in this research, except that they can choose which mattress they want to lie on. Additionally, participation can help us gain more knowledge to make radiotherapy treatment more comfortable. Participation in the research will not affect the treatment. Participants will receive the normal treatment and check-ups for their condition. The drawback of participating is that the investigators will ask patients to try both mattresses, which will take about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 16
* Patients treated for bone metastasis in thoracic, abdominal and pelvic region
* Patients have read, understood and signed the informed consent of the COMFORT study (in Dutch).

Exclusion Criteria:

* Patients not willing or able to test two mattresses (RT-Comfort Mattress and standard thin foam matt)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
The percentage of patients that prefered the newly developed comfort mattress over the standard thin foam matt | Prior to radiotherapy planning-CT acquisition.
  The included patients tested the RT-Comfort Mattress and standard thin foam matt by lying on each for one minute in radiotherapy position, on the flat and hard CT scanner couch. Next, after patients identified their mattress or matt of choice, the treatment preparation and delivery were performed on their mattress or matt of choice according to standard clinical practice.

SECONDARY OUTCOMES:
The level preferrence of patients for the mattress of choice. | Prior to radiotherapy planning-CT acquisition.
  The included patients tested the regular matt and the RT-Comfort Mattress by lying on each for one minute in radiotherapy position, on the flat and hard CT scanner couch. Next, they identified their mattress of choice, and the level of preference; slight or strong.
The pain patients experienced while lying on the comfort mattress and the standard thin foam matt, according to the 11-point Numerical Rating Scale (NRS). | Prior to radiotherapy planning-CT acquisition, while lying on each mattress for one minute in treatment position.
  The 11-point NRS ranges from 0 (equivalent to no pain) to 10 (the worst pain imaginable).
The positioning stability of patients on the comfort mattress and the standard thin foam matt, measured with optical surface scanning | During the first treatment fraction, the patients' surface scanning measurements were started directly after CBCT positioning verification and stopped directly after treatment dose delivery.
  The positioning stability on the mattress was considered sufficient if two requirements were met; (1) the sagging (i.e.: the change in vertical position over time) during the first 5 minutes of dose delivery should be less than 1 mm averaged over all patients, (2) the variation in vertical position over time should not be larger compared to patients positioned during treatment on the standard matt.
The dosimetrical effect of the RT-Comfort Mattress in the beam | The dosimetrical effect was evaluated immediately after the radiotherapy treatment.
  As negligible dosimetric effect was expected, the original treatment plan was generated in the treatment planning system without taking the RT-Comfort mattress in account. To investigate the expected negligible effect of the mattress attenuation on 95% dose coverage of the planning target volume (PTV) and maximum skin dose, the treatment plans were recalculated and reoptimized while accounting for the RT-Comfort mattress using the same treatment planning system. The skin contour was defined as the outer 5-mm of the patient body contour for all CT-slices that included a PTV contour. The PTV itself was excluded from the skin structure.

CONTACTS AND LOCATIONS:
Overall Officials: Remi Nout, Proffessor, Study Director — Erasmus MC Cancer Institute
Locations (1):
- Erasmus MC Cancer Institute, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
According to the IRB approved study protocol, collected data will not be exchanged, shared or transferred outside the Erasmus MC. All data is handled conform the Dutch Act on Implementation of the General Data Protection Regulation (in Dutch: Uitvoeringswet Algemene Verordening Gegevensbescherming (UAVG)) and the Erasmus MC privacy regulations. For sharing of data with other parties patients need to be informed and they should agree for that as part of the informed consent procedure. The patients included in this study did not provide written informed consent for sharing of their data with other parties as data sharing with others was not included in the patient information folder.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT06903507/Prot_SAP_000.pdf